CLINICAL TRIAL: NCT07047781
Title: Relationship Between Smartphone Addiction and Thoracic Hyperkyphosis in Children
Brief Title: Smartphone Addiction and Thoracic Hyperkyphosis in Children
Status: Completed | Type: Observational
Sponsor: Istinye University (Other)
Responsible Party: Principal Investigator, Kubra Koce, Asst. Prof., Istinye University
Other Study IDs: 23/114
Record Dates: First submitted 2025-06-23; First posted 2025-07-02 (Actual); Last update posted 2025-08-21 (Actual); Status verified 2025-08

CONDITIONS: Hyperkyphosis
Keywords: smartphone addiction; thoracic hyperkyphosis; posture
MeSH Terms: conditions — Kyphosis; Internet Addiction Disorder | interventions — Restraint, Physical

STUDY DESIGN:
Observational Model: Other | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (1):
- Group 1: Individuals between the ages of 7 and 14 who are receiving primary education and meet the inclusion criteria will be included in this study planned to evaluate the relationship between smartphone addiction and thoracic hyperkyphosis in children with thoracic hyperkyphosis.
  Interventions: Other: Assessment

INTERVENTIONS:
Other: Assessment — Individuals between the ages of 7 and 14 who are receiving primary education and meet the inclusion criteria will be included in this study planned to evaluate the relationship between smartphone addiction and thoracic hyperkyphosis in children with thoracic hyperkyphosis.

SUMMARY:
Smartphones are advanced devices that have evolved beyond basic calling and messaging functions, offering features comparable to computers due to the development of mobile operating systems. In addition to their technical capabilities, smartphones have become increasingly appealing to children, adolescents, and adults through continuously updated websites, applications, and social networks that provide access to current information and opportunities for social interaction.

Excessive use of smartphones and similar technological devices can be defined as mobile phone addiction or internet addiction. The risk of smartphone addiction is particularly high among children and adolescents. The prolonged use of smartphones, which are now an integral part of daily life, may negatively affect physical capacity, including the musculoskeletal system. Previous studies have shown that increased smartphone use is associated with neck/shoulder and upper extremity/back discomfort. This increased usage can lead to non-neutral spinal postures and sustained muscular loading. Due to the central role of the spine within the kinetic chain, postural changes and muscular strain in the spine may affect movement quality in both upper and lower segments. For example, excessive neck flexion while texting can have widespread effects on spinal alignment and function. Therefore, smartphone use may cause significant changes in thoracic kyphosis and lumbar lordosis.

Thoracic hyperkyphosis is commonly detected during adolescence and encompasses a range of spinal deformities from mild postural changes to rigid deformities accompanied by soft tissue and structural alterations. In children and adolescents, three main types of hyperkyphosis are observed: postural kyphosis, Scheuermann's kyphosis, and congenital kyphosis.

Postural hyperkyphosis is the most common type. It results from the weakness of antigravity muscles responsible for upright posture, leading to curvature of the spine under external forces. This type of curvature is not rigid and can often be corrected voluntarily when the individual is instructed to stand upright. Postural hyperkyphosis typically occurs during adolescence and is characterized by a thoracic kyphosis angle generally below 65 degrees. It is a common yet often overlooked condition in healthy adolescents and can be identified through school screenings.

Today, the growing use of smartphones and the associated rise in technology addiction have contributed to the increasing prevalence of postural hyperkyphosis, which is caused by prolonged incorrect postures. It has also been reported that postural habits developed during childhood often persist into adulthood.

If left untreated, hyperkyphosis that begins in adolescence may continue into adulthood, potentially increasing healthcare expenditures. With the rising incidence of hyperkyphosis linked to smartphone addiction, it is crucial to address this deformity beginning in adolescence, both from a health and economic perspective. Many authorities advocate for the inclusion of scoliosis and hyperkyphosis in school screening programs. However, routine screenings for skeletal system problems are not conducted in schools. Moreover, the limited number of studies in this area have primarily focused on scoliosis, and to date, no screening studies have addressed hyperkyphosis specifically.

ELIGIBILITY:
Inclusion Criteria:

* Being between 7-14 years old
* Using a smartphone for more than a year
* Daily smartphone usage time >60 minutes

Exclusion Criteria:

* Those who have had major surgery or trauma related to the musculoskeletal system, especially the spine and upper extremities
* Difficulty in perceiving commands
* Rigid deformity in the spine (Scheuermann Kyphosis)
* Congenital deformity

Ages: 7 Years to 14 Years | Sex: All
Age Groups: Child
Study Population: Individuals between the ages of 7 and 14 who are receiving primary education and meet the inclusion criteria will be included in this study planned to evaluate the relationship between smartphone addiction and thoracic hyperkyphosis in children with thoracic hyperkyphosis.
Sampling Method: Probability Sample
Enrollment: 77 (Actual)
Dates: Start 2025-06-23 (Actual); Primary Completion 2025-08-01 (Actual); Study Completion 2025-08-01 (Actual)

PRIMARY OUTCOMES:
Sociodemographic Status Assessment | 4 weeks
  The sociodemographic status of the participants will be recorded with an assessment form prepared by the researchers. Information on age, gender, dominant side, duration and habits of smartphone use,will be questioned. Participants' privacy will be respected throughout the study, and no photographs will be taken.
Smartphone Addiction Scale-Short Form | 4 weeks
  Smartphone Addiction Scale-Short Form will be used to measure smartphone addiction. The smartphone addiction scale, developed to measure the risk of smartphone addiction in young people, is a six-point Likert-type scale consisting of 10 items with one factor (1: strongly disagree and 6: strongly 15 agree) and is based on self-reporting. The internal consistency and concurrent validity of the scale were confirmed with a Cronbach's alpha of 0.911. The total score is minimum 10 and maximum 60. It was evaluated that the risk of addiction increases as the score increases. In the Korean sample, the cut-off value was specified as 31 for men and 33 for women. Turkish validity and reliability studies were conducted by Noyan et al. in 2014.
Flexicurve Ruler | 4 weeks
  Flexicurve Ruler will measure thoracic curvature and calculate kyphosis index. Kyphosis index is the value found by dividing the width of the thoracic curvature by its length.
Wall-Occiput Distance | 4 weeks
  The increase in the thoracic kyphosis angle will be evaluated and recorded with the wall-occiput distance measurement. The distance between the occiput and the wall will be measured with a ruler while the individual to be tested is standing in contact with the wall.
Posture analysis with Posture Screen Mobile Application | 4 weeks
  Posture analysis will be used to determine postural deviations that may occur in individuals. Posture analysis will be performed via the "Posture Screen" application, which can be accessed via smartphones.
Range of Motion | 4 weeks
  Cervical region flexion, extension, lateral flexion and rotation movements, upper extremity shoulder flexion, extension movements, trunk flexion, lateral flexion and extension angles will be measured bilaterally with a digital goniometer. Measurements will be repeated 3 times and the average value will be recorded in degrees
The shortness of the pectoral muscles | 4 weeks
  The shortness of the pectoral muscles will be evaluated with a tape measure.
Sit-Reach test | 4 weeks
  The shortness of the hamstring muscle will be evaluated with the Sit-Reach test.
Satisfaction with Body Image | 4 weeks
  There is no scale specific to hyperkyphosis deformity in the literature that evaluates individuals' perception of satisfaction with their body image. In the existing studies in the literature, a numerical scale between 0 and 10 was used to evaluate how the perception of satisfaction with body image changes in hyperkyphosis deformity. According to the scale, 0 represents very satisfied with appearance, while 10 represents not satisfied with appearance at all.
Height | 4 weeks
  The vertical distance from the top of the head to the heels of the individual. It will be measured in centimeters.
Weight | 4 weeks
  The mass of the individual's body in relation to gravity. It will be expressed in kilograms.
Waist Circumference | 4 weeks
  A circumferential measurement taken with a tape measure at the narrowest point of the waist, or at the midpoint between the lower margin of the last palpable rib and the top of the iliac crest, to assess abdominal fat distribution. It will be measured in centimeters.

CONTACTS AND LOCATIONS:
Locations (1):
- Istinye University, Istanbul, Turkey (Türkiye)

IPD SHARING:
Plan to Share IPD: Undecided